CLINICAL TRIAL: NCT06241482
Title: A Randomized Controlled Clinical Study on Safety and Efficacy of Enhanced Recovery After Surgery in Neurocritical Care Patients
Brief Title: Safety and Efficacy of Enhanced Recovery After Surgery in Neurocritical Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hao Chen, MD, PhD, Associate Professor, Chief Physician, Graduate Supervisor, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-179
Record Dates: First submitted 2024-01-20; First posted 2024-02-05 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Neurocritical Care; Traumatic Brain Injury; Cerebrovascular Disease; Moderate or Severe Coma
Keywords: Neurocritical Care; Traumatic Brain Injury; Cerebrovascular Disease
MeSH Terms: conditions — Brain Injuries, Traumatic; Cerebrovascular Disorders; Lymphoma, Follicular; Coma | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced recovery after surgery (Experimental): The technologies, processes and measures of enhanced recovery after surgery were applied.
  Interventions: Procedure: Enhanced recovery after surgery
- Conventional therapy (Active Comparator): Conventional therapy were applied.
  Interventions: Procedure: Conventional therapy

INTERVENTIONS:
Procedure: Enhanced recovery after surgery — The technologies, processes and measures of enhanced recovery after surgery focus on the following aspects:
  1. Early assessment and treatment
  2. Optimized anesthetic protocol
  3. Reducing surgical stress
  4. Multi-modal comprehensive monitoring
  5. Comprehensive diagnosis and treatment in neurosurgical intensive care
  6. Intensive early rehabilitation treatment
  Arms: Enhanced recovery after surgery
Procedure: Conventional therapy — Conventional therapy in neurocritical care.
  Arms: Conventional therapy

SUMMARY:
Enhanced recovery after surgery (ERAS) is a strategy of perioperative management aimed to accelerate the rehabilitation of patients through various optimized perioperative managements as well as ongoing adherence to a patient-focused, multidisciplinary, and multimodal approach. Alleviating the injury and stress caused by surgery or disease is the core principle of ERAS, which has been shown to reduce complication rates after surgery, promote patient recovery, decrease hospital length of stay and reduce costs. ERAS has been widely applied in many surgical perioperative fields, and it has achieved remarkable effects. However, there are few applications of ERAS in neurosurgery, especially in clinical trials of neurocritical care patients.

Therefore, the investigators attempt to conduct the study of ERAS in neurosurgical intensive patients using a series of optimized perioperative managements that have been verified to be effective by evidence-based medicine, and to evaluate the safety and effectiveness of ERAS in neurocritical care. The aim of this study is to explore the most suitable ERAS protocols to accelerate the postoperative rehabilitation process of neurocritical care patients, and to provide more evidence-based medicine for the effectiveness and safety of ERAS in neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old
* Patients with moderate or severe acute traumatic brain injury or cerebrovascular disease requiring neurosurgical intensive care treatment
* Hospitalization time ≥ 1 week
* The guardian is able to understand and actively cooperate in completing the project
* The guardian signs an informed consent form

Exclusion Criteria:

* Patients undergoing non-surgical treatment
* Patients diagnosed as brain death within the first 24 hours after admission to NICU
* Patients undergoing cardiopulmonary resuscitation, maintenance dialysis, end-stage tumors, and disseminated cancer
* Patients who withdraw treatment during hospitalization or are discharged automatically
* Patients who underwent unplanned secondary surgery during the research process
* Individuals who cannot be followed up during the research process

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Clinical prognosis | One month, three and six months after injury or attack
  Glasgow Outcome Scale score (1 = death; 2 = persistent vegetative state; 3 = severe disability; 4 = moderate disability; 5 = good but not necessarily complete recovery; unfavorable outcome was defined as score of ≤3, and favorable outcome was defined as a score of >3)
Neurological function assessment | One month, three and six months after injury or attack
  Modified Rankin scale score (0 = no symptoms; 1 = no significant disability; 2 = slight disability; 3 = moderate disability; 4 = moderately severe disability; 5 = severe disability; 6 = dead; favorable outcome was defined as score of 0-2, and unfavorable outcome was defined as score of 3-6)

SECONDARY OUTCOMES:
Neuroimaging evaluation | One week, two weeks after surgery; one month, three and six months after injury or attack
  Computer tomography or magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Hao Chen, M.D., Ph.D., Study Director — Shanghai 6th Peoples' Hospital
Locations (1):
- Shanghai 6th People's Hospital, Shanghai, China